CLINICAL TRIAL: NCT04381156
Title: The Involvement of microRNAs in the Recovery From Acute Kidney Injury
Brief Title: MicroRNAs in Renal Recovery - Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, PD Dr. Timo Brandenburger, Principal Investigator, Heinrich-Heine University, Duesseldorf
Other Study IDs: 6138
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Markers in Plasma and Urine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this Pilot study, the potential of noncoding RNAs in renal recovery from acute kidney injury will be evaluated.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in almost 50% of patients treated in intensive care units. AKI mainly occurs after sepsis, acute ischemia, nephrotoxicity or hypoxia and leads to severe damage of the kidney and to an increased risk of mortality. The diagnosis of AKI is currently based on creatinine, urea and diuresis. Yet, novel markers may improve the accuracy of this diagnosis at an early stage of the disease, thereby allowing for early prevention and therapy, ultimately leading to a reduction of the need for renal replacement therapy and decreased mortality. Several potential biomarkers have been examined in the context of AKI in the last years [e. g. Cystatin C, a cysteine protease inhibitor, NGAL (neutrophil gelatinase-associated lipocalin), KIM-1 (kidney injury molecule 1), and IGFBP7 (insulin like growth factor binding protein 7) and TIMP-2 (tissue inhibitor of metalloproteinase 2)].

These biomarkers may help to identify AKI earlier and more reliable in the future.

However, recovery of renal function during/after AKI is not predictable with the classical biomarkers creatinine and urea. Only a few studies have analyzed the potential of several new biomarkers in the prediction of renal recovery during AKI including urinary hepatocyte growth factor (uHGF), urinary IGFBP- 7 and TIMP-2 or NGAL. Still, their ability to predict renal recovery remains unclear and in clinical practice, recovery of renal function is estimated empirically including the decision to discontinue renal replacement therapy. In a consensus statement from 2017 on behalf of the Acute Disease Quality Initiative Workgroup 16 it is stated that more research is needed to "determine optimal methods to assess functional recovery and identify novel biomarker(s) [...] that can inform ongoing injury and repair in AKD".

In the ncRNA in renal recovery study we therefore aim to analyze the potential of microRNAs (miRNAs) and circular RNA (circRNAs) in predicting recovery of renal function in critically ill patients suffering from AKI. Non-coding RNAs emerged during the past few years as important regulatory molecules that allow a fine-tuning of gene expression and protein synthesis. This regulation is necessary to maintain homeostasis and its dysregulation is often associated with disease development. Non-coding RNAs are present in the kidney and in body fluids and their expression is modulated during AKI and their potential as biomarkers in various diseases has been shown. As ncRNAs are involved in injury and repair of kidneys, they may represent an interesting class of molecules with a potential as biomarkers and therapeutic targets in recovery from AKI.

Blood and urine samples will be collected at 4 different time points (day 0, day 1, day 2 and day 7). Plasma miRNAs will be screened for differential miRNA expression by next generation sequencing (5 patients with early recovery versus 5 patients with no signs of recovery). Differentially expressed miRNAs will then be analyzed by qPCR in plasma and urine.

The proposed study is aimed to better understand the pathophysiological basis of recovery from AKI and may form the basis of further studies for biomarker and therapeutics research in renal recovery.

ELIGIBILITY:
Inclusion Criteria:

* AKI stage 2 or 3

Exclusion Criteria:

* kidney transplantation
* eGFR < 30 ml/Min
* dialysis within last 90 days
* chronic dialysis
* pregnancy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with AKI
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of ncRNAs as markers in renal recovery from AKI | 1 yr
  Observation

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesiologie, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided